CLINICAL TRIAL: NCT07031908
Title: Minimally Invasive Interval Debulking Surgery in Advanced Ovarian Cancer, a Prospective Observational Study
Brief Title: Minimally Invasive Interval Debulking Surgery in Advanced Ovarian Cancer
Acronym: MISSION-2
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7596
Record Dates: First submitted 2025-06-04; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Minimally invasive cytoreduction — Minimally invasive cytoreduction in patients with advanced ovarian cancer treated with 6 cycles of neoadjuvant chemotherpy

SUMMARY:
In women with advanced epithelial ovarian cancer (AOC), neoadjuvant chemotherapy (NACT) combined with interval cytoreductive surgery and post-operative chemotherapy is an option.

Several retrospective studies have demonstrated the feasibility of minimally invasive surgery in case of a good response to neoadjuvant chemotherapy, and prospective randomised trial is currently underway to demonstrate the non-inferiority of minimally invasive surgery compared to laparotomy in patients with an optimal response after 3-4 cycles of neoadjuvant chemotherapy (LANCE trial, NCT04575935).

The aim of our study is to evaluate the feasibility of interval surgery after at least VI cycles of neoadjuvant chemotherapy with a minimally invasive approach.

DETAILED DESCRIPTION:
In women with advanced epithelial ovarian cancer (AOC), neoadjuvant chemotherapy (NACT) combined with interval cytoreductive surgery (ICS) and post-operative chemotherapy is an option. Four randomised trials (EORTC55971, CHORUS, JCOG0602, SCORPION) have shown that survival rates after NACT are similar to those after primary cytoreductive surgery and adjuvant chemotherapy.

The use of neoadjuvant chemotherapy has increased significantly in recent years, and it has been shown that the determining prognostic factor is the achievement of an absent residual tumour at surgery. However, the optimal number of neoadjuvant chemotherapy cycles is not yet well defined. Several retrospective studies have evaluated the efficacy of interval debulking surgery after performing more than 4 cycles of neoadjuvant chemotherapy. In these studies, the percentage of patients undergoing >4 cycles of neoadjuvant chemotherapy varied in a range of approximately 22% to 45%. Currently, several randomised trials are ongoing, evaluating the optimal number of neoadjuvant chemotherapy cycles (3 vs. 6 cycles) in terms of complete cytoreduction (GOGER, NCT02125513) and survival (CHRONO, NCT03579394).

Several retrospective studies have demonstrated the feasibility of minimally invasive surgery in case of a good response to neoadjuvant chemotherapy (median neoadjuvant chemotherapy cycles: 4). Therefore, a prospective randomised trial is currently underway to demonstrate the non-inferiority in terms of progression-free survival of minimally invasive surgery compared to laparotomy in patients with an optimal response after 3-4 cycles of neoadjuvant chemotherapy (LANCE trial, NCT04575935).

The aim of our study is to evaluate the feasibility of interval surgery after at least VI cycles of neoadjuvant chemotherapy with a minimally invasive approach.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIC or IV high-grade invasive epithelial ovarian carcinoma (serous, endometrioid, clear cell, transitional), primary peritoneal carcinoma, or fallopian tube carcinoma, or pathology consistent with high-grade Müllerian carcinoma.
* Partial or complete radiological response of abdominal cavity disease after at least 6 cycles of neoadjuvant chemotherapy (NACT).
* CA125 < 100 U/mL.
* ECOG performance status 0-1.
* Signed informed consent and ability to comply with follow-up, including in cases where the patient has a legal guardian. In such cases, consent will be provided by the legal guardian.
* Review of imaging by a radiologist and senior surgeon at a multidisciplinary tumor board, particularly evaluating hepatic hilum involvement, mesenteric root, extensive peritoneal disease in the upper abdomen, extensive hepatic or gastric involvement, and extensive intestinal involvement.
* If all the previous criteria are met and protocol acceptance is obtained, the patient will undergo a laparoscopic evaluation of all abdominal quadrants to confirm the feasibility of minimally invasive surgery (MIS). Surgery will be considered feasible if complete gross resection can be achieved with minimally invasive surgery. If minimally invasive surgery is not feasible, the patient will be excluded from the study, and the reason for unfeasibility will be described.

Exclusion Criteria:

* Evidence of a tumor not amenable to minimally invasive complete resection on preoperative imaging (CT, PET-CT, or MRI). Radiologic criteria (tumor board evaluation): hepatic hilum involvement, mesentery root, extensive peritoneal disease in upper abdomen, extensive hepatic or gastric involvement, extensive intestinal involvement
* Disease free of other active malignancies within the past 5 years, except basal cell carcinoma of the skin.
* History of psychological, familial, sociological, or geographic conditions potentially impeding adherence to the study protocol and follow-up program
* Inability to tolerate prolonged Trendelenburg position or pneumoperitoneum

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with primary advanced epithelial ovarian cancer, FIGO stage III-IV not candidate for primary debulking surgery at diagnosis or after III-IV cycles of neoadjuvant chemotherapy.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2029-06-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of minimally invasive surgery | 15 days
  Minimally invasive surgery feasibility will be calculated on the rates of: conversion from MIS to laparotomy, complete gross resection, and protocol acceptance. In this study feasibility is defined as a conversion rate <20%, a complete gross resection rate >80% and the enrollment of at least 1 patient each month.
Safety of minimally invasive surgery (First parameter) | 2 years
  2 Years Overall Survival defined as the interval time (months) between surgery and death or censored at the last follow-up
Safety of minimally invasive surgery (Second parameter) | 2 years
  2 Years Disease Free Survival defined as the interval time (months) between surgery and the first occurrence of relapse or death due to ovarian cancer, whichever occurs first or censored at the last follow-up
Safety of minimally invasive surgery (third parameter) | 6 months
  Safety will be evaluated using the following criteria:
  - Rate of early and late severe post-operative complications (early: <30days from surgery; late: more than 30 days and less then 6 months from surgery) using Clavien Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Conte, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, UOC Ginecologia Oncologica, Roma, Italy